CLINICAL TRIAL: NCT00948818
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial of Linaclotide Administered Orally for 12 Weeks Followed by a 4-Week Randomized Withdrawal Period in Patients With Irritable Bowel Syndrome With Constipation
Brief Title: Trial of Linaclotide Administered to Patients With Irritable Bowel Syndrome With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-31
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
Keywords: Irritable Bowel Syndrome; Constipation; Linaclotide
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linaclotide (Experimental): Linaclotide 290 micrograms
  Interventions: Drug: Linaclotide 290 micrograms
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Linaclotide 290 micrograms — Oral, once daily each morning at least 30 minutes before breakfast for the duration of the study
  Arms: Linaclotide
Drug: Matching placebo — Oral, once daily each morning at least 30 minutes before breakfast for the duration of the study
  Arms: Placebo

SUMMARY:
The objective of this trial is to determine the efficacy and safety of linaclotide administered to patients with irritable bowel syndrome with constipation (IBS-C).

The primary efficacy parameter is the percentage of patients in each treatment group that meet the protocol definition for Abdominal Pain and Complete Spontaneous Bowel Movement (APC) Responder.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets protocol criteria for IBS: reports abdominal discomfort or pain that has two or more of the following three features:

  1. Relieved with defecation
  2. Onset associated with a change in frequency of stool
  3. Onset associated with a change in form (appearance) of stool
* Patient reports < 3 bowel movements (BMs) per week (in the absence of any laxative, suppository, or enema use during the preceding 24 hours) and reports straining, lumpy or hard stools, and/or sensation of incomplete evacuation during > 25% of BMs
* Patient has successfully completed protocol procedures (with no clinically significant findings): physical exam, 12-lead ECG, or clinical laboratory tests (some patients may require a colonoscopy per American Gastroenterological Association (AGA) guidelines)
* Patient is compliant with Interactive Voice Response System (IVRS) for daily diary reporting of BM habits and IBS symptoms

Exclusion Criteria:

* Patient has history of loose or watery stools for >25% of BMs
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a history of a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history or concomitant medication use that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F.C. Eng, PhD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (118):
- United States (111):
  - Forest Investigative Site 037, Birmingham, Alabama
  - Forest Investigative Site 036, Birmingham, Alabama
  - Forest Investigative Site 135, Hueytown, Alabama
  - Forest Investigative Site 014, Huntsville, Alabama
  - Forest Investigative Site 080, Chandler, Arizona
  - Forest Investigative Site 053, Mesa, Arizona
  - Forest Investigative Site 078, Peoria, Arizona
  - Forest Investigative Site 101, Phoenix, Arizona
  - Forest Investigative Site 128, Phoenix, Arizona
  - Forest Investigative Site 051, Scottsdale, Arizona
  - Forest Investigative Site 136, Tucson, Arizona
  - Forest Investigative Site 087, Tucson, Arizona
  - Forest Investigative Site 094, Burbank, California
  - Forest Investigative Site 026, Encinitas, California
  - Forest Investigative Site 096, Foothill Ranch, California
  - Forest Investigative Site 057, Los Angeles, California
  - Forest Investigative Site 097, Mission Hills, California
  - Forest Investigative Site 005, Orange, California
  - Forest Investigative Site 024, Westlake Village, California
  - Forest Investigative Site 021, Boulder, Colorado
  - Forest Investigative Site 019, Colorado Springs, Colorado
  - Forest Investigative Site 034, Denver, Colorado
  - Forest Investigative Site 074, Longmont, Colorado
  - Forest Investigative Site 010, Wheat Ridge, Colorado
  - Forest Investigative Site 058, Waterbury, Connecticut
  - Forest Investigative Site 042, Boca Raton, Florida
  - Forest Investigative Site 003, Bradenton, Florida
  - Forest Investigative Site 137, Brandon, Florida
  - Forest Investigative Site 070, Brooksville, Florida
  - Forest Investigative Site 018, Fort Myers, Florida
  - Forest Investigative Site 030, Jupiter, Florida
  - Forest Investigative Site 077, Kissimmee, Florida
  - Forest Investigative Site 133, Miami, Florida
  - Forest Investigative Site 031, Miami, Florida
  - Forest Investigative Site 129, New Smyrna Beach, Florida
  - Forest Investigative Site 108, Ocala, Florida
  - Forest Investigative Site 092, Orlando, Florida
  - Forest Investigative Site 038, Panama City, Florida
  - Forest Investigative Site 027, Pembroke Pines, Florida
  - Forest Investigative Site 045, St. Petersburg, Florida
  - Forest Investigative Site 015, Tampa, Florida
  - Forest Investigative Site 104, Trinity, Florida
  - Forest Investigative Site 068, Zephyrhills, Florida
  - Forest Investigative Site 032, Atlanta, Georgia
  - Forest Investigative Site 103, Atlanta, Georgia
  - Forest Investigative Site 033, Marietta, Georgia
  - Forest Investigative Site 020, Marietta, Georgia
  - Forest Investigative Site 040, Woodstock, Georgia
  - Forest Investigative Site 055, Idaho Falls, Idaho
  - Forest Investigative Site 043, Rockford, Illinois
  - Forest Investigative Site 047, Evansville, Indiana
  - Forest Investigative Site 046, Iowa City, Iowa
  - Forest Investigative Site 029, Arkansas City, Kansas
  - Forest Investigative Site 009, Newton, Kansas
  - Forest Investigative Site 023, Wichita, Kansas
  - Forest Investigative Site 093, Wichita, Kansas
  - Forest Investigative Site 067, Lexington, Kentucky
  - Forest Investigative Site 114, Madisonville, Kentucky
  - Forest Investigative Site 132, Baton Rouge, Louisiana
  - Forest Investigative Site 124, Shreveport, Louisiana
  - Forest Investigative Site 013, Chevy Chase, Maryland
  - Forest Investigative Site 006, Hagerstown, Maryland
  - Forest Investigative Site 073, Lutherville, Maryland
  - Forest Investigative Site 001, Boston, Massachusetts
  - Forest Investigative Site 125, Kalamazoo, Michigan
  - Forest Investigative Site 064, Chaska, Minnesota
  - Forest Investigative Site 004, St Louis, Missouri
  - Forest Investigative Site 085, Vineland, New Jersey
  - Forest Investigative Site 052, Albuquerque, New Mexico
  - Forest Investigative Site 035, Brooklyn, New York
  - Forest Investigative Site 017, Great Neck, New York
  - Forest Investigative Site 011, Great Neck, New York
  - Forest Investigative Site 134, Setauket, New York
  - Forest Investigative Site 122, Boone, North Carolina
  - Forest Investigative Site 072, Fayetteville, North Carolina
  - Forest Investigative Site 016, Greensboro, North Carolina
  - Forest Investigative Site 119, Hickory, North Carolina
  - Forest Investigative Site 088, Raleigh, North Carolina
  - Forest Investigative Site 056, Wilmington, North Carolina
  - Forest Investigative Site 065, Winston-Salem, North Carolina
  - Forest Investigative Site 028, Cincinnati, Ohio
  - Forest Investigative Site 044, Cleveland, Ohio
  - Forest Investigative Site 123, Columbus, Ohio
  - Forest Investigative Site 130, Dayton, Ohio
  - Forest Investigative Site 082, Oklahoma City, Oklahoma
  - Forest Investigative Site 102, Tulsa, Oklahoma
  - Forest Investigative Site 039, Pittsburgh, Pennsylvania
  - Forest Investigative Site 121, Greenville, South Carolina
  - Forest Investigative Site 069, Greer, South Carolina
  - Forest Investigative Site 131, Greer, South Carolina
  - Forest Investigative Site 025, Nashville, Tennessee
  - Forest Investigative Site 099, Austin, Texas
  - Forest Investigative Site 002, Dallas, Texas
  - Forest Investigative Site 041, Houston, Texas
  - Forest Investigative Site 110, Houston, Texas
  - Forest Investigative Site 063, Lake Jackson, Texas
  - Forest Investigative Site 095, San Antonio, Texas
  - Forest Investigative Site 076, San Antonio, Texas
  - Forest Investigative Site 089, Salt Lake City, Utah
  - Forest Investigative Site 091, Salt Lake City, Utah
  - Forest Investigative Site 100, Salt Lake City, Utah
  - Forest Investigative Site 054, Charlottesville, Virginia
  - Forest Investigative Site 061, Christianburg, Virginia
  - Forest Investigative Site 007, Newport News, Virginia
  - Forest Investigative Site 060, Norfolk, Virginia
  - Forest Investigative Site 075, Norfolk, Virginia
  - Forest Investigative Site 050, Richmond, Virginia
  - Forest Investigative Site 049, Bellevue, Washington
  - Forest Investigative Site 098, Lakewood, Washington
  - Forest Investigative Site 066, Wenatchee, Washington
  - Forest Investigative Site 083, Milwaukee, Wisconsin
- Canada (7):
  - Forest Investigative Site 113, Greater Sudbury, Ontario
  - Forest Investigative Site 107, Hamilton, Ontario
  - Forest Investigative Site 112, Newmarket, Ontario
  - Forest Investigative Site 106, Ottawa, Ontario
  - Forest Investigative Site 115, Sarnia, Ontario
  - Forest Investigative Site 008, Toronto, Ontario
  - Forest Investigative Site 116, Toronto, Ontario

REFERENCES:
- [Derived] Rao SS, Quigley EM, Shiff SJ, Lavins BJ, Kurtz CB, MacDougall JE, Currie MG, Johnston JM. Effect of linaclotide on severe abdominal symptoms in patients with irritable bowel syndrome with constipation. Clin Gastroenterol Hepatol. 2014 Apr;12(4):616-23. doi: 10.1016/j.cgh.2013.09.022. Epub 2013 Sep 25. PMID 24075889
- [Derived] Quigley EM, Tack J, Chey WD, Rao SS, Fortea J, Falques M, Diaz C, Shiff SJ, Currie MG, Johnston JM. Randomised clinical trials: linaclotide phase 3 studies in IBS-C - a prespecified further analysis based on European Medicines Agency-specified endpoints. Aliment Pharmacol Ther. 2013 Jan;37(1):49-61. doi: 10.1111/apt.12123. Epub 2012 Nov 1. PMID 23116208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over an eight month period from July 2009 to March 2009 at 118 study sites (111 in the United States, 7 in Canada).
Pre-assignment Details: Patients went through a 14 to 21 day Pretreatment Period during which the patients provided qualifying bowel habit and symptoms, and rescue medicine usage information through an interactive voice response system (IVRS). All randomized patients needed an abdominal pain score ≥ 3. One randomized patient in the Placebo arm did not receive study drug.
Groups:
- Placebo: Dose-matched placebo, oral administration, once per day.
- Linaclotide: Linaclotide 290µg, oral administration, once per day.
Period: Overall Study
Arm/Group | Placebo | Linaclotide
Started | 397 | 406
Completed | 335 | 312
Not Completed | 62 | 94
Not completed — Adverse Event | 10 | 32
Not completed — Protocol Violation | 9 | 10
Not completed — Withdrawal by Subject | 25 | 25
Not completed — Lost to Follow-up | 10 | 17
Not completed — Lack of Efficacy | 4 | 5
Not completed — Other Reason | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide | Total
Number analyzed (Participants) | 396 | 406 | 802
Age Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.9) | 43.3 (12.7) | 43.5 (12.8)
Age, Customized [Number; unit: participants]
  18 years to 64 years | 370 | 387 | 757
  65 years and older | 26 | 19 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358 | 368 | 726
  Male | 38 | 38 | 76
Region of Enrollment [Number; unit: participants]
  United States | 367 | 374 | 741
  Canada | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Abdominal Pain and Complete Spontaneous Bowel Movement (APC) Responder, 9 Out of 12 Weeks
Description: A patient is considered to be an APC responder if, for at least 9 out of the 12 weeks of the treatment period, the patient had at least 3 CSBMs, experienced an increase of at least 1 CSBM from baseline, and experienced a decrease of at least 30 percent in their Abdominal Pain (AP) score from baseline during a particular week.
  The AP score assesses the worst of a patient's AP in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no AP and 10 represents very severe AP.
  A CSBM is defined as a spontaneous bowel movement, associated with a sense of complete evacuation.
Time Frame: Change from Baseline to Week 12
Population: 803 patients were randomized to treatment, and 802 patients received double-blind study drug. 800 patients had at least 1 postrandomization entry of the primary efficacy assessment and were included in the Intent to Treat (ITT) Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Number; unit: Participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Participants
  Responder | 20 | 49
  Nonresponder | 375 | 356
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 9/12 Week APC 3 + 1 Responders. The power, adjusted for multiplicity, was expected to be 93% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — The p-value is still less than 0.05 after adjusting multiplicity using a serial gatekeeping multiple comparison procedure; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.51 to 4.47]

2. Secondary Outcome: 12-Week Complete Spontaneous Bowel Movement (CSBM) Frequency Rate
Description: The number of CSBMs per week.
Time Frame: Change from Baseline to Week 12
Population: 803 patients were randomized to treatment, and 802 patients received double-blind study drug. 800 patients had at least 1 postrandomization entry of the primary efficacy assessment and were included in the ITT Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: CSBMs per Week
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
CSBMs per Week | 0.705 (0.128) | 2.272 (0.127)

3. Primary Outcome: Complete Spontaneous Bowel Movement (CSBM) 3+1 Responder, 9 Out of 12 Weeks
Description: A patient is considered to be a CSBM 3+1 responder if, for at least 9 out of the 12 weeks of the treatment period, the patient had at least 3 CSBMs and experienced an increase of at least 1 CSBM from baseline during a particular week.
  A CSBM was defined as a Spontaneous Bowel Movement (SBM) that was associated with a sense of complete evacuation.
  An SBM was defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: Participant
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Participant
  Responder | 25 | 79
  Non-responder | 370 | 326
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 9/12 Week CSBM 3 + 1 Responders. The power, adjusted for multiplicity, was expected to be 93% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.65, 95% CI 2-sided [2.26 to 5.88]

4. Primary Outcome: Abdominal Pain Responder, 9 Out of 12 Weeks
Description: A patient is considered to be an abdominal pain responder if, for at least 9 out of the 12 weeks of the treatment period, they experienced a decrease of at least 30 percent in the mean abdominal pain score from baseline during a particular week.
  The Abdominal Pain score assesses the worst of a patient's abdominal pain in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Participants
  Responder | 107 | 139
  Non-responder | 288 | 266
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 9/12 Week Abdominal Pain Responders. The power, adjusted for multiplicity, was expected to be 93% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p = 0.0262, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.04 to 1.91]

5. Primary Outcome: Abdominal Pain and Complete Spontaneous Bowel Movement (APC) Responder, 6 Out of 12 Weeks.
Description: A patient is considered an APC responder if, for at least 6 of the 12 weeks of the treatment, the patient experienced an increase of at least 1 Complete Spontaneous Bowel Movement (CSBM) from baseline and experienced a decrease of at least 30 percent in their Abdominal Pain (AP)score during a particular week.
  The AP score assesses the worst of a patient's AP in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no AP and 10 represents very severe AP.
  A CSBM was defined as a Spontaneous Bowel Movement (SBM) that was associated with a sense of complete evacuation.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Participants
  Responder | 83 | 136
  Non-responder | 312 | 269
Statistical Analysis 1: Comparison: Placebo vs Linaclotide; Null Hypothesis: There is no difference between the 290 μg dose and placebo groups in the proportion of 6/12 Week APC + 1 Responders. The power, adjusted for multiplicity, was expected to be 86% based on NCT00460811 (MCP-103-202) study data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.40 to 2.66]

6. Secondary Outcome: 12-Week Spontaneous Bowl Movement (SBM) Frequency Rate
Description: The number of Spontaneous Bowl Movements experienced per week.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
SBMs per week | 1.130 (.0177) | 3.898 (0.176)

7. Secondary Outcome: 12-Week Stool Consistency
Description: The consistency of each BM was assessed by patients using the 7-point Bristol Stool Form Scale (BSFS) from 1 to 7.
  1. = separate hard lumps like nuts [difficult to pass]
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges [passed easily]
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces [entirely liquid]).
Time Frame: Change from Baseline to Week 12
Population: 802 randomized patients received study drug. The 800 patients in the ITT population had at least 1 postrandomization entry of the primary efficacy assessment; 107 patients with no pretreatment spontaneous bowel movements were excluded from the 12-Week Stool Consistency analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 338 | 355
units on a scale | 0.662 (0.061) | 2.071 (0.060)

8. Secondary Outcome: 12-Week Severity of Straining
Description: Straining is measured on a 5-point scale where a value of 1 is "not at all" and a value of 5 is "an extreme amount.
Time Frame: Change from Baseline to Week 12
Population: 802 randomized patients received study drug. The 800 patients in the ITT population had at least 1 postrandomization entry of the primary efficacy assessment; 107 patients with no pretreatment spontaneous bowel movements were excluded from the Severity of Straining analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 338 | 355
units on a scale | -0.651 (0.042) | -1.306 (0.042)

9. Secondary Outcome: 12-Week Change in Abdominal Pain Score
Description: Abdominal Pain at its worst (in the last 24 hours) is based on an 11-point scale where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
units on a scale | -1.129 (0.094) | -1.869 (0.093)

10. Secondary Outcome: 12-Week Change in Abdominal Discomfort
Description: Abdominal Discomfort is measured on an 11-point scale where a value of 0 is "none" and a value of 10 is "very severe."
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
units on a scale | -1.211 (0.097) | -1.953 (0.096)

11. Secondary Outcome: 12-Week Change in Bloating
Description: Bloating was assessed on an 11-point scale where a value of 0 is "none" and a value of 10 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
units on a scale | -1.100 (0.100) | -1.944 (0.099)

12. Secondary Outcome: Complete Spontaneous Bowl Movement (CSBM) Responder for 6 Weeks Out of 12 Weeks of Treatment
Description: A patient is considered to be a CSBM responder if, for at least 6 out of the 12 weeks of the treatment period, an increase of at least 1 CSBM per week from baseline was experienced.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Participants
  Responder | 117 | 197
  Non-responder | 278 | 208

13. Secondary Outcome: Abdominal Pain Responder for 6 Out of 12 Weeks
Description: A patient is considered to be an abdominal pain responder if, for at least 6 out of the 12 weeks of the treatment period, they experienced a decrease of 30 percent or more in the abdominal pain score from baseline.
  The Abdominal Pain score assesses the worst of a patient's abdominal pain in the past 24 hours using an 11-point scale (from 0-10), where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Participants
  Responder | 148 | 203
  Non-Responder | 247 | 202

14. Secondary Outcome: 12-Week Percent of Abdominal Pain-free (APF) Days
Description: Abdominal pain free (APF) days are those days where the patient reported a score of '0' for abdominal pain at its worst
  Abdominal Pain at its worst (in the last 24 hours) is based on an 11-point scale where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Linaclotide
Number analyzed (Participants) | 395 | 405
Percent | 5.31 (15.74) | 9.81 (21.75)

ADVERSE EVENTS:
Time Frame: Adverse event data for the treatment period was collected from July of 2009 to July of 2010
Description: 803 patients were randomized to treatment. A total of 802 patients received double-blind study drug and were included in the Safety Population.
Groups:
- Placebo - Treatment Period: Dose-matched placebo, oral administration, once per day.
- Linaclotide - Treatment Period: Linaclotide 290µg, oral administration, once per day.
- Placebo to Linaclotide - Randomized Withdrawal Period: Linaclotide 290µg, oral administration, once per day during a 4-week randomized withdrawal period.
  This group had previously received dose-matched placebo during the 12-week randomized treatment period.
- Linaclotide to Placebo - Randomized Withdrawal Period: Dose-matched placebo, oral administration, once per day during a 4-week randomized withdrawal period.
  This group had previously received linaclotide 290µg, oral administration, once per day during the 12-week treatment period.
- Linaclotide to Linaclotide - Randomized Withdrawal Period: Linaclotide 290µg, oral administration, once per day during a 4-week randomized withdrawal period
Arm/Group | Placebo - Treatment Period | Linaclotide - Treatment Period | Placebo to Linaclotide - Randomized Withdrawal Period | Linaclotide to Placebo - Randomized Withdrawal Period | Linaclotide to Linaclotide - Randomized Withdrawal Period
Serious Adverse Events (participants affected / at risk) | 2/396 | 2/406 | 0/333 | 0/154 | 0/158
Other Adverse Events (participants affected / at risk) | 22/396 | 93/406 | 41/333 | 1/154 | 5/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Treatment Period (N=396) | Linaclotide - Treatment Period (N=406) | Placebo to Linaclotide - Randomized Withdrawal Period (N=333) | Linaclotide to Placebo - Randomized Withdrawal Period (N=154) | Linaclotide to Linaclotide - Randomized Withdrawal Period (N=158)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Treatment Period (N=396) | Linaclotide - Treatment Period (N=406) | Placebo to Linaclotide - Randomized Withdrawal Period (N=333) | Linaclotide to Placebo - Randomized Withdrawal Period (N=154) | Linaclotide to Linaclotide - Randomized Withdrawal Period (N=158)
Diarrhea (General disorders) | 14 | 79 | 39 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 10 | 22 | 8 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this trial will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the trial. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.